CLINICAL TRIAL: NCT07168915
Title: A Randomized, Double-Blind Study to Evaluate the Safety, Tolerability, and Immunogenicity of V118 Formulation E in Healthy Adults
Brief Title: A Study of V118E in Healthy Participants (V118E-003)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: V118E-003
Record Dates: First submitted 2025-09-04; First posted 2025-09-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Healthy
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- V118E (Experimental): Participants receive intramuscular (IM) injection of V118E in a 2-dose regimen administered on Day 1 and Day 29.
  Interventions: Biological: V118E
- PREVNAR 20™ + Saline (Active Comparator): Participants receive one dose of IM injection of PREVNAR 20™ in a 2-dose regimen on Day 1 followed by one dose of saline on Day 29.
  Interventions: Biological: PREVNAR 20™; Biological: Saline

INTERVENTIONS:
Biological: V118E — IM administration
  Other Names: V118/VA-017
  Arms: V118E
Biological: PREVNAR 20™ — IM administration
  Arms: PREVNAR 20™ + Saline
Biological: Saline — IM administration
  Arms: PREVNAR 20™ + Saline

SUMMARY:
Researchers are looking for new vaccines to prevent illnesses caused by a type of bacteria called Streptococcus pneumoniae. There are many different types of Streptococcus pneumoniae bacteria, called serotypes. Vaccines contain small parts of certain serotypes. These parts will not cause an infection but help the body create antibodies (proteins) to fight the bacteria.

PREVNAR 20™ is a vaccine given to help to prevent disease from Streptococcus pneumoniae bacteria. Researchers designed a new vaccine, V118E, to help prevent disease from Streptococcus pneumoniae bacteria.

The goal of this study is to learn how safe V118 formulation E is in Healthy Adults and how well people tolerate it.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

- Is in good health before randomization

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has a history of invasive pneumococcal disease or known history of other culture-positive pneumococcal disease within 3 years prior to receiving study vaccination
* Has a history of clinically significant endocrine, gastrointestinal (GI), cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2027-05-10 (Estimated); Study Completion 2027-05-10 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Solicited Injection-Site Adverse Events (AEs) | Up to approximately 7 days after each vaccination
  An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, which occurs during the course of the study. A solicited AE is a predefined event that participants are specifically asked about and record on their vaccine report card (VRC). Solicited injection-site AEs include redness, swelling, and pain or tenderness. The number of participants with a solicited injection-site AE will be reported.
Number of Participants With Solicited Systemic AEs | Up to approximately 7 days after each vaccination
  An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, which occurs during the course of the study. A solicited AE is a predefined event that participants are specifically asked about and record on their VRC. Solicited systemic AEs include fever, muscle aches all over body, joint pain, headache, and tiredness. The number of participants with a solicited systemic AE will be reported.
Number of Participants With Immediate AEs Following Vaccination | Up to approximately 30 minutes after each vaccination
  An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, which occurs during the course of the study. The number of participants with immediate AEs following vaccination will be reported.
Number of Participants With Unsolicited AEs | Up to approximately 28 days after each vaccination
  An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, which occurs during the course of the study. An unsolicited AE is an event that is not solicited using a VRC and that is communicated by a participant. The number of participants who experience an unsolicited AE will be reported.
Number of Participants With a Serious Adverse Event (SAE) | Up to approximately 12 months after final vaccination
  An SAE is defined as any untoward medical occurrence that at any dose, results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect. The number of participants who experience an SAE will be reported.
Number of Participants With a Medically Attended Adverse Event (MAAE) | Up to approximately 12 months after final vaccination
  A MAAE is defined as an adverse event in which medical attention is received during an unscheduled, non-routine outpatient visit, such as an emergency department visit, office visit, or an urgent care visit with any medical personnel for any reason. The number of participants who experience a MAAE will be reported.
Number of Participants With an Adverse Events of Special Interest (AESI) | Up to approximately 12 months after final vaccination
  AESIs are selected serious and nonserious AEs which include but are not limited to: 1) Potential drug-induced liver injury (DILI) events defined as an elevated aspartate aminotransferase (AST) or alanine aminotransferase (ALT) laboratory value that is ≥3* the upper limit of normal (ULN) and an elevated total bilirubin laboratory value that is ≥2* the ULN and, at the same time, an alkaline phosphatase laboratory value that is <2* the ULN, as determined by way of protocol-specified laboratory testing or unscheduled laboratory testing. 2) an overdose of V118E. 3) Potential immune-mediated disease (pIMDs) defined as a subset of AEs that an established autoimmune disease(s) AND inflammatory and/or neurologic disorder(s), which might or might not have an autoimmune etiology. The number of participants who experience an AESI will be reported.

SECONDARY OUTCOMES:
Serotype-specific Immunoglobulin G (IgG) Geometric Mean Concentrations (GMCs) | Day 28 Postvaccination 1
  The GMCs for serotype-specific IgG antibodies will be determined using pneumococcal electrochemiluminescence (Pn ECL) assay.
Change From Baseline in Serotype-specific IgG GMCs | Baseline and Day 28 Postvaccination 1
  Change from baseline in GMCs for serotype-specific IgG antibodies will be determined using Pn ECL assay.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (4):
- United States (4):
  - Velocity Clinical Research, Hallandale Beach ( Site 0003), Hallandale, Florida
  - QPS-MRA, LLC-Early Phase ( Site 0002), South Miami, Florida
  - Bio-Kinetic Clinical Applications, LLC dba QPS-MO ( Site 0004), Springfield, Missouri
  - University of Texas Medical Branch ( Site 0001), Galveston, Texas

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com